CLINICAL TRIAL: NCT04127448
Title: Effect of Virtual Reality Based Exercise Training v/s Aerobic Exercises on Cognitive Function in Adults With Type 2 Diabetes Mellitus.
Brief Title: Exergaming Versus Aerobic Exercises on Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah IU Raana Ali
Record Dates: First submitted 2019-09-25; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes; Cognitive Impairment
Keywords: Aerobic Exercise; Cognitive dysfunction; Exergaming; T2DM.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming Training Group (Experimental): Training was given using X-box 360 Kinect.
  Interventions: Other: Exergaming Training Group
- Aerobic Exercise Group (Active Comparator): Session using treadmill (model no TMX58 220).
  Interventions: Other: Aerobic Exercise Group

INTERVENTIONS:
Other: Exergaming Training Group — Training was given using X-box 360 Kinect. Dr. Kawashima's brain and body exercise game comprising of multiple cognitive games out of which 4 selected games were played by the participants. These games were "Traffic control" (participants have to guide the colored cars into their matching colored tunnels by using their arms), "balloon buster" (players pop numbered balloons in order from the lowest to the highest), "pop till u drop", (match the color that appears on screen with the balloon of same color) and "strike a pose" (participant have to remember the poses shown and then copy them after few seconds). Games were played for 10 minutes initially then the duration was gradually increased to 30 minutes each session for 3 days/week and duration of 6 weeks. The session included 5-minute warm up, 20-minute interactive gaming, and 5-minute cool down.
  Arms: Exergaming Training Group
Other: Aerobic Exercise Group — Session of 30-35 minutes, 3 days a week for 6 weeks was given using treadmill (model no TMX58 220). Time and intensity was gradually increased over the duration of 6 weeks. Starting from 10 minutes in 1st week, every 5 minutes was added to aerobics phase to each week until patient reached to 35 minutes in week 6 maintaining the intensity of 40-60% of heart rate reserve (%HRR).
  Arms: Aerobic Exercise Group

SUMMARY:
The ain to this study was to determine the effects of Exergaming and Aerobic exercise on mild cognitive impairment (MCI) and random blood sugar levels (RBS) in adults with type 2 diabetes mellitus (T2DM) and to compare the effects between both treatments.This Randomized Control Trial (RCT) enrolled 33 diabetics to Aerobic group (AG) (n=18) and Exergaming training group (ER) (n=15) who completed the six weeks of aerobics or ER training. Aerobic group followed intervention using treadmill for 30 mins/day for 3 days/week maintaining intensity of 40-60% heart rate reserve (HRR). The ER group did physical activity using X-box 360 for 30 mins/day, 3 days/week. The cognitive testing included MMSE, MOCA, Trail-A/B and verbal fluency test (VF). The random blood sugar levels (RBS) of the participants were also monitored. Data was analyzed on IBM SPSS Statistics 20.

DETAILED DESCRIPTION:
The American Diabetes Association define diabetes as a metabolic disorder characterized by decreased production of insulin and/or the development of insulin resistance which results in hyperglycemia. The most common types of DM are type 1 and type 2. Type 2 diabetes mellitus (T2DM) is more commonly observed in adults and represents 90-95% cases worldwide. According to WHO, Pakistan is ranked 7th among countries with high prevalence rate of T2DM. A review done in December 2016 stated that the prevalence rate of T2DM in Pakistan is 11.77%. (Males =11.20% /females=9.19%).

Diabetes mellitus is found to be associated with a vast majority of co-morbidities that have devastating impact on the health and quality of life of the patients. Among diabetics the development of cardiovascular dysfunctions is a well known cause of mortality and morbidity. Around 80% diabetic populations develop the metabolic syndrome, characterized by the development of insulin resistance along with hypertension, Dyslipidemia and visceral obesity. Obesity is very commonly observed among diabetics and the occurrence of visceral adiposity contributes to the increment of the pathogenesis of insulin resistance. Other co-morbidities associated with diabetes are diabetic retinopathy, neuropathy, nephropathy, psychosocial impairments and cognitive dysfunction.

It is well known that diabetes mellitus is found to be associated with many co-morbidities. Recent evidences show that it is also a risk factor for the development of cognitive impairment. Studies show that diabetics have a 1.2- to 1.5-fold greater rate of developing decline in cognitive function compared to those without diabetes. A 15 year follow up study done in Japan in 2011 also reported increased prevalence of dementia among the diabetics. It is becoming evident that diabetes affects the nervous system causing diabetic encephalopathy which results in the neuronal damage and loss contributing to cognitive dysfunction. A review published in 2009 stated that mild to moderate cognitive declines were observed among diabetics. Reduced performance was observed on the tests of multiple cognitive domains including episodic memory, information processing speeds and task executive functioning. A little decline was also observed on the tests concerning mental flexibility. It is becoming evident from the data of epidemiological studies that there is strong association between diabetes and increased risk of pathological changes in central nervous system resulting in cognitive dysfunction and later on developing into dementia. A review states that it is evident from the neurocognitive testing that cognitive decline should be listed among the many diabetes associated complications. The factors like the end organ damage influenced by hyperglycemia, vascular and neuronal damage, hypoglycemia and the presence of amyloid lesions may be held responsible for the changes and damages to cerebral structure. Literature shows that cognitive dysfunction is also related with the diabetes associated co-morbidities including Increased obesity, Low muscle mass, depression, cardiovascular diseases, chronic inflammation and cerebrovascular diseases.

Diet and exercise represent the initial treatment approaches in clinical practice to slow progression of metabolic disturbance associated with prediabetes and to assist with pharmacological treatment in established T2DM. Increased physical activity has clear beneficial physiological effects for older adults with T2DM or glucose intolerance or insulin resistance and more recently has been shown to benefit cognition as well.Epidemiological evidence consistently links physical exercise with better cognitive performance, lower risks for dementia, and reduced pathological changes in the central nervous system (CNS). Experimental studies have also reported benefits of aerobic and resistance training on cognitive function in older adults.

The trend towards using the virtual reality as a platform for rehabilitation among many neurological deficits is increasing tremendously. Researches show that VR training may be helpful in improving the physical, cognitive and emotional impairments faced by the patients experiencing some neurological deficit. It has been seen that when patients following brain insult after stroke are involved in VR related rehabilitation programs their functional performance was improved. The improvements were seen in balance, walking speeds and mobility.

Although no trials have been done to our knowledge concerning the use of virtual reality and cognitive dysfunctions in adults with T2DM but a variety of researches indicate that VR can be useful in treating cognitive impairments. Undoubtedly VR training has potential to simulate many real life or imaginary situations, hence providing the platform for more valid and dynamic assessment and training. It also provides a constant environment with the prospective for multiple repetitions of the same task to be assessed. Furthermore in contrast to many conventional methods, VR-based assessment and training provides accurate performance measurements and exact replays of task performance. Currently VR is being used as a supportive intervention after brain damage to deal with multiple aspects of cognitive impairments including memory impairment, executive dysfunctions, visio-spatial and attention deficit. The use of VR brain damage rehabilitation is exceedingly expanding and will become an important part of cognitive assessment and rehabilitation in future. Studies also show VR as a beneficial tool for treating anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* subjects scoring <25 on MMSE
* subjects being treated with diet alone, oral medications, insulin or combination at the time of enrolment, without recent changes in medication (<3 months)
* sedentary adults (self-reporting of < 30 min of structured physical activity for < 3 times/week during last 6 months)

Exclusion Criteria:

* if they had any co-morbidity that presented contraindications to moderate to vigorous type of physical activity.
* Subjects with any unstable chronic diseases or significant cognitive impairment (diagnosed dementia) were also excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Standardized Mini-mental State Examination (SMMSE) from baseline to 6th week. | The score were recorded at baseline before intervention start and at the 6th week i.e. at the end of intervention.
  Among diabetics it is an effective tool for the assessment of global cognition. It is a 30 points questionnaire with 20 separate tests. The twenty individual tests consist of eleven main areas of construction, writing, orientation, attention, registration, calculation, repetition, recalls. Scores of less then 25 are considered as person having impaired cognition.
Change in Montreal cognitive assessment scale (MOCA, Urdu version) from baseline to 6th week. | The score were recorded at baseline before intervention start and at the 6th week i.e. at the end of intervention.
  It is a 30-point test administered in approximately 10 minutes. Thirty items assessing multiple cognitive domains include short-term memory, executive function, verbal ability, visuospatial abilities, sustained-attention task etc. The scores of less the 26 are considered to be abnormal.
Change in Trail Making Test-A (TMT-A) from baseline to 6th week | The score were recorded at baseline before intervention start and at the 6th week i.e. at the end of intervention.
  Twenty-five circles are distributed over a piece of paper, and the circles enclose a number ranging from 1 to 25. Subjects are asked to connect the circles in numerical sequence as quickly and accurately as possible without lifting their pencil from the paper.
Change in Trail Making Test-B (TMT-B) from baseline to 6th week | The score were recorded at baseline before intervention start and at the 6th week i.e. at the end of intervention.
  Trail making Test-B (TMT-B): There are 25 circles with numbers from 1 to 12 along with 12 Urdu alphabets in them. Participants are required to connect the circles in an alternating progressive sequence as quickly and accurately as possible without lifting their pencil from the paper. Trail-B is a pure test of assessing the executive functioning.
Change in Verbal fluency test (VFT) from baseline to 6th week | The score were recorded at baseline before intervention start and at the 6th week i.e. at the end of intervention.
  It is a test to assess the verbal ability and executive control ability. It consists of 2 tasks: semantic fluency and phonemic fluency and the participants are given 1 min to produce as many unique words as possible within these categories. In semantic category participants have to produce name of objects for example fruits or animals. In phonemic words starting from a specific letter like 'f' are produced. The participant's score in each task is the number of unique correct words.

SECONDARY OUTCOMES:
Change in Random Blood sugar (RBS) from baseline to 6th week | The score were recorded for 6 weeks before the start of each session.
  Blood sugar (RBS) was measured using glucometer (ACCU-CHECK Performa, model= NC (mg/dl) Sr no: 68802207857) before each session.

OTHER OUTCOMES:
Change in Blood pressure in mm Hg from baseline to 6 week | The score were recorded for 6 weeks before and after each session.
  Blood pressure was monitored before and after each session. Mercury Sphagmomanometer and Stethoscope was used to monitor blood pressure.
Change in pulse rate in beats/min from baseline to 6 week | The score were recorded for 6 weeks before and after each session.
  Pulse rate was monitored before and after each session. Cardiac monitor (Operon OM-12) was used to monitor pulse rate and O2 sat. Cardiac monitor (Operon OM-12) was used to monitor pulse rate.
Change in oxygen saturation (O2 sat) in percentage from baseline to 6th week. | The score were recorded for 6 weeks before and after each session.
  Oxygen saturation (O2 sat) was monitored before and after each session. Cardiac monitor (Operon OM-12) was used to monitor pulse rate and O2 sat. Cardiac monitor (Operon OM-12) was used to monitor Oxygen saturation.
Change in respiratory rate in breaths/min from baseline to 6th week. | The score were recorded for 6 weeks before and after each session.
  Respiratory rate was monitored before and after each session. Respiratory was measured through abdominal movements in supine lying.

CONTACTS AND LOCATIONS:
Overall Officials: Irum Yaqoob, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Standards of medical care in diabetes-2015 abridged for primary care providers. Clin Diabetes. 2015 Apr;33(2):97-111. doi: 10.2337/diaclin.33.2.97. No abstract available. PMID 25897193
- [Background] Meo SA, Zia I, Bukhari IA, Arain SA. Type 2 diabetes mellitus in Pakistan: Current prevalence and future forecast. J Pak Med Assoc. 2016 Dec;66(12):1637-1642. PMID 27924966
- [Background] Greenberg AS, Obin MS. Obesity and the role of adipose tissue in inflammation and metabolism. Am J Clin Nutr. 2006 Feb;83(2):461S-465S. doi: 10.1093/ajcn/83.2.461S. PMID 16470013
- [Background] Cukierman T, Gerstein HC, Williamson JD. Cognitive decline and dementia in diabetes--systematic overview of prospective observational studies. Diabetologia. 2005 Dec;48(12):2460-9. doi: 10.1007/s00125-005-0023-4. Epub 2005 Nov 8. PMID 16283246
- [Background] Luchsinger JA. Type 2 diabetes and cognitive impairment: linking mechanisms. J Alzheimers Dis. 2012;30 Suppl 2(0):S185-98. doi: 10.3233/JAD-2012-111433. PMID 22433668
- [Background] S Roriz-Filho J, Sa-Roriz TM, Rosset I, Camozzato AL, Santos AC, Chaves ML, Moriguti JC, Roriz-Cruz M. (Pre)diabetes, brain aging, and cognition. Biochim Biophys Acta. 2009 May;1792(5):432-43. doi: 10.1016/j.bbadis.2008.12.003. Epub 2008 Dec 16. PMID 19135149
- [Background] Roberts RO, Geda YE, Knopman DS, Christianson TJ, Pankratz VS, Boeve BF, Vella A, Rocca WA, Petersen RC. Association of duration and severity of diabetes mellitus with mild cognitive impairment. Arch Neurol. 2008 Aug;65(8):1066-73. doi: 10.1001/archneur.65.8.1066. PMID 18695056
- [Background] Kodl CT, Seaquist ER. Cognitive dysfunction and diabetes mellitus. Endocr Rev. 2008 Jun;29(4):494-511. doi: 10.1210/er.2007-0034. Epub 2008 Apr 24. PMID 18436709
- [Background] Awad N, Gagnon M, Messier C. The relationship between impaired glucose tolerance, type 2 diabetes, and cognitive function. J Clin Exp Neuropsychol. 2004 Nov;26(8):1044-80. doi: 10.1080/13803390490514875. PMID 15590460
- [Background] Kawamura T, Umemura T, Hotta N. Cognitive impairment in diabetic patients: Can diabetic control prevent cognitive decline? J Diabetes Investig. 2012 Oct 18;3(5):413-23. doi: 10.1111/j.2040-1124.2012.00234.x. Epub 2012 Aug 29. PMID 24843599
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Suzuki T, Shimada H, Makizako H, Doi T, Yoshida D, Tsutsumimoto K, Anan Y, Uemura K, Lee S, Park H. Effects of multicomponent exercise on cognitive function in older adults with amnestic mild cognitive impairment: a randomized controlled trial. BMC Neurol. 2012 Oct 31;12:128. doi: 10.1186/1471-2377-12-128. PMID 23113898
- [Background] Nagamatsu LS, Handy TC, Hsu CL, Voss M, Liu-Ambrose T. Resistance training promotes cognitive and functional brain plasticity in seniors with probable mild cognitive impairment. Arch Intern Med. 2012 Apr 23;172(8):666-8. doi: 10.1001/archinternmed.2012.379. No abstract available. PMID 22529236
- [Background] Rose FD, Brooks BM, Rizzo AA. Virtual reality in brain damage rehabilitation: review. Cyberpsychol Behav. 2005 Jun;8(3):241-62; discussion 263-71. doi: 10.1089/cpb.2005.8.241. PMID 15971974
- [Background] Corbetta D, Imeri F, Gatti R. Rehabilitation that incorporates virtual reality is more effective than standard rehabilitation for improving walking speed, balance and mobility after stroke: a systematic review. J Physiother. 2015 Jul;61(3):117-24. doi: 10.1016/j.jphys.2015.05.017. Epub 2015 Jun 18. PMID 26093805